CLINICAL TRIAL: NCT06565546
Title: Feasibility and Efficacy of CYP2D6 Genotype-guided Management of Opioid Analgesics in Patients Undergoing Elective Ventral Hernia Repairs: A Pilot Pragmatic Trial
Brief Title: CYP2D6 Genotype-guided Management of Opioid Analgesics in Patients Undergoing Elective Ventral Hernia Repairs
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 202401069
Record Dates: First submitted 2024-08-13; First posted 2024-08-22 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-03

CONDITIONS: Ventral Hernia
MeSH Terms: conditions — Hernia, Ventral | interventions — Acetaminophen; Gabapentin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CYP2D6 genotype testing-treatment (Experimental): CYP2D6 genotype testing performed preoperatively with results used to guide prescribing of opioid analgesics during the postoperative period to control pain. In addition, participants will receive standard of care postoperative pain medications.
  Interventions: Other: Opioid pain medication prescribed based on CYP2D6 genotype testing PLUS Acetaminophen and Gabapentin
- CYP2D6 genotype testing-control (Active Comparator): CYP2D6 genotype testing performed preoperatively, results will be delayed until after operative procedure. Participants will receive standard of care postoperative pain medication prescriptions for pain management.
  Interventions: Other: Acetaminophen and Gabapentin: standard postoperative pain medications

INTERVENTIONS:
Other: Opioid pain medication prescribed based on CYP2D6 genotype testing PLUS Acetaminophen and Gabapentin — CYP2D6 genotype testing for assessment of medication metabolism to guide prescription of postoperative pain medication
  Arms: CYP2D6 genotype testing-treatment
Other: Acetaminophen and Gabapentin: standard postoperative pain medications — Participants will receive standard postoperative pain medications
  Arms: CYP2D6 genotype testing-control

SUMMARY:
Pilot pragmatic trial using an implementation science approach to determine the feasibility of a CYP2D6-guided opioid prescribing for patients undergoing elective VHRs compared to usual care. Assess the efficacy (PROMIS Pain Intensity and Hernia-Related QOL) of a CYP2D6-guided opioid prescribing approach for patients undergoing elective VHRs.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years age undergoing a ventral hernia repair (VHR) ≥1.5 cm in diameter with mesh.

Exclusion Criteria:

* ventral hernia <1.5 cm
* primary ventral hernia repair (VHR) without a mesh
* emergency operative procedure
* receiving chronic opioid therapy (defined as use of opioids on most days for >3 months)
* allergy to opioids
* women of childbearing potential who have a positive pregnancy result as part of their standard pre-surgical workup

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-01-29 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Determine the feasibility of a CYP2D6-guided opioid prescribing by the percentage enrolled of patients undergoing elective VHRs compared to usual care. | 6 months
  Percentage of potential participants approached will enroll and complete study.

SECONDARY OUTCOMES:
Assess the efficacy of a CYP2D6-guided opioid prescribing approach for patients undergoing elective VHRs. | 6 months
  Participants may report improved post-operative pain control and quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Jana Sacco, MD, Principal Investigator — Assistant Professor
Locations (1):
- University of Florida Jacksonville, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No